CLINICAL TRIAL: NCT05315674
Title: Early Diagnostic BioMARKers in Exacerbations of COPD: the MARKED Study
Brief Title: Markers of COPD Exacerbations
Acronym: MARKED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Center of Expertise for Chronic Organ Failure (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Frits M. E. Franssen, Principal Investigator, Center of Expertise for Chronic Organ Failure
Other Study IDs: MARKED
Record Dates: First submitted 2022-03-08; First posted 2022-04-07 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: COPD; COPD Exacerbation
Keywords: COPD; COPD Exacerbation; Microbiota; Biomarker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biosamples of spontaneous sputum, the nasopharynx, venous blood and stool will be frequently collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exacerbators: Patients who experience ≥1 inpatient AECOPD
  Interventions: Diagnostic Test: Frequent assessment of biomarker panel
- Non-exacerbators: Patients without inpatient AECOPD
  Interventions: Diagnostic Test: Frequent assessment of biomarker panel

INTERVENTIONS:
Diagnostic Test: Frequent assessment of biomarker panel — During the eight-week inpatient follow-up period there will be daily follow-up of respiratory symptoms, vitals and spirometry, and a thrice weekly collection of spontaneous sputum, nasal swabs and venous blood. These assessments will be repeated at acute worsening of respiratory symptoms at which a stool sample will also be collected.

SUMMARY:
Acute exacerbations of COPD (AECOPD) are episodes of acute worsening of respiratory symptoms that require additional therapy. Exacerbations play a pivotal role in the burden and progressive course of COPD (1). Each event contributes to a progressive decline in lung function (2), reduced health status, low physical activity level (3) and increased health care costs (4). As such, disease management is predominantly based on the prevention of these episodes (1). Yet, in the Netherlands, 30.000 people are admitted to the hospital for an AECOPD every year (5). Although most AECOPD have an infectious origin (6), the underlying mechanisms are heterogeneous and predicting their occurrence in individual patients currently remains unsuccessful (7-9). Furthermore, there is a lack of our understanding in the longitudinal alterations in microbial composition and host-microbiome interactions in the stable state, at AECOPD and during recovery in patients with COPD. This knowledge is essential to improve the early and accurate diagnosis of (the different types of) AECOPD, and for the development of novel antimicrobial and other therapeutic targets and subsequent personalized treatment. These challenges need to be addressed in order to reduce the future impact of these events, avoid unnecessary treatments of individual patients, reduce healthcare utilization and improve overall care for patients with COPD. The current 'Early diagnostic BioMARKers in Exacerbations of COPD' (MARKED) study was designed to investigate several of these gaps in the management of COPD exacerbations.

It is anticipated that complex biomarker panels, rather than a single biomarker, will be identified. Since AECOPD are heterogeneous events in terms of origin, trigger, severity, duration, need for treatment and overall clinical presentation (1, 6, 10-15), we expect to identify different biomarker panels for different subtypes of AECOPD. Furthermore, AECOPD diagnosis relies heavily on the exclusion of differential diagnoses (1), which further rules out the potential of a single predictive AECOPD biomarker.

DETAILED DESCRIPTION:
The MARKED study is an exploratory, prospective, single-center, longitudinal, observational study with eight weeks follow-up. The primary objective is to explore which biomarkers from a panel of frequently measured biomarkers (symptoms, vital signs, lung function parameters and spontaneous sputum, nasopharyngeal swabs, stool and blood samples) predict an exacerbation and/or respiratory infection in patients with COPD. Furthermore, secondary objectives are:

I. to investigate longitudinal alterations in microbial composition and host-microbiome interactions in the stable state, at AECOPD and during recovery.

II. to study the heterogeneity of AECOPD by comprehensive clinical, functional, microbial, proteomic, transcriptomic, genetic, metabolomic, inflammatory and biochemical characterization of these events.

III. to determine the correlation between microbial alterations in the airways/gut and inflammatory biomarkers in blood during longitudinal follow up.

IV. to longitudinally investigate biomarkers of AECOPD in clinically relevant subgroups of patients with COPD (e.g. current versus ex-smokers, high versus low blood eosinophils, frequent vs. infrequent exacerbators).

V. to comprehensively investigate whether host-microbiome interactions, biomarkers and predictive models identify those patients that do not exacerbate despite having a respiratory infection.

All AECOPD evaluated by the physician in Ciro as moderate or severe will be recorded in this study. Moderate AECOPD are defined by a worsening of symptoms >2 consecutive days leading to treatment with systemic glucocorticoids, antibiotics or both. Severe events are characterized by (enhanced) oxygen therapy, non-invasive ventilation (NIV) or hospital admission that lasted >24 hours, in addition to treatment with systemic glucocorticoids, antibiotics or both.

Whilst aiming to include at least 50 patients experiencing an AECOPD and at least 50 patients without an AECOPD, up to 150 consecutive patients with a primary diagnosis of COPD admitted for inpatient pulmonary rehabilitation at Ciro will be recruited for the study. Although sample size rules of thumb exist for multivariable regression modelling and prediction modelling strategies, this study is explorative in nature. Therefore, the amount of biomarkers exceeds the amount when applying the rule of thumb that states that for each potential predictive variable, 10 events should be observed. The study aims to include at least 50 unique individual patients who experience ≥1 AECOPD, and at least 50 individual patients without an AECOPD, to provide accurate benchmark data (i.e. sufficient precision to estimate mean and standard deviation [SD]) for exploratory biomarkers. From previous studies in Ciro it is known that approximately 42% of patients will develop at least one AECOPD during admission (16). Because AECOPD are unpredictable and variable, which is an important rationale for the present study, the study will expectedly need 100-150 patients to be included. The goal of this study is not to develop a multivariate model, but rather to explore the associations between biomarkers and the occurrence of an event.

Baseline characteristics will be reported as mean and SD or as median and interquartile range (IQR) for continuous variables, as appropriate, and as count and percentage for categorical characteristics. Predictors of time-to-first AECOPD during the study period will be modelled using univariate and multivariable Cox proportional hazards regression. Associations will be presented as hazard ratio (HR) and 95% confidence interval (CI). The dependency of the predictive performance of biomarkers will be tested using interaction terms. The concordance-statistic, or c-statistic, will be estimated to assess discriminative ability. Time-dependent AUC-Receiver Operating Characteristics (ROC) plots will furthermore be created. Calibration will be assessed by comparing the predicted probability with the observed probability of an AECOPD, and examined with a calibration plot and calibration slope, assuming no data censoring before the end of follow-up.

Characterization of the microbiome will be determined by alpha- and beta-diversity and relative abundance of bacterial taxa. Alpha-diversity will be treated as a continuous variable and analysed using appropriate statistical tests, whereas ordination of beta-diversity distances will be done using principal component analysis. Multiomic analyses will be used to generate hypotheses about the drivers that promote progression to AECOPD. Differential enrichment analysis for feature selection across all 'omics will be done after accounting for multiple hypothesis testing using a robust model that considers distributional assumptions. The association between genetic variants and (AE)COPD and microbial infections will be studied using whole-exome sequencing data.

Self-organizing maps (SOMs, also referred to as Kohonen maps) will be used to create an ordered representation of the selected attributes at the time of AECOPD by using Viscovery Profiler 7.1 (Viscovery Software GmbH, Vienna, Austria). Based on the identified homogeneous data groups created in the SOM model, clusters will be generated using Viscovery's SOM-Ward Cluster algorithm. Summary variables of clinical characteristics for the total sample, and for clusters, will be presented as mean and SD for quantitative variables, and as percentages for discrete variables. Differences between groups will be assessed using integrated two-sided t-tests. Repeated measure correlations will be used to determine the within-individual association between microbial alterations in the airways/gut and systemic inflammatory biomarkers across patients.

In case of missing data on predictors, stochastic regression imputation with fully conditional specification will be used to impute the dataset to allow the use of all included patients for the analyses. Values will be drawn using predictive mean matching. Statistical significance will be denoted by p<0.05.

The current study is classified as research with negligible risk. There are no serious risks associated with participation in this study. Hematomas might occur from venous blood sampling. Nasal discomfort might be experienced during nasal sampling. Patients might experience breathlessness and fatigue due to additional daily measurements (e.g. questionnaires, lung function) and/or might refuse participation or drop-out of the study because of the burden of frequent sampling and other assessments. Extensive guidelines have been established to monitor scientific research in a structured and protocol-based manner at Ciro. In the context of the NFU report 'Quality assurance for people-related research', the current investigator initiated research was classified as research with negligible risk. The assigned study site monitor will monitor the safety of the participants, and the accuracy of following procedures as described in the protocol by the research staff, on an annual basis. Monitoring will be performed in compliance with Good Clinical Practice (GCP) in order to achieve high quality research and secure patient safety.

In accordance with the Medical Research Involving Human Subjects Act (WMO) the study will be suspended if the health or safety of subjects will be jeopardised. The accredited Medical Ethical Teaching Committee (Medical Research Ethics Committees United [MEC-U], Nieuwegein, the Netherlands) will be notified without undue delay after obtaining knowledge of these events. Adverse and serious adverse events will be recorded. Hospitalized AECOPD will not be considered as serious adverse events. Exacerbations and hospitalized AECOPD will be annually reported to MEC-U. Ciro has established protocols for the management of AECOPD; these protocols will also be followed for patients included in the study. Moderate AECOPD are treated at Ciro, the pulmonary rehabilitation program will be adjusted as needed. Patients with severe AECOPD requiring hospital admission will be referred to a nearby hospital.

Ethical approval for the study has been granted by MEC-U (NL71364.100.19). The study will be conducted according to the principles of the Declaration of Helsinki (64th WMA General Assembly, Fortaleza, Brazil, October 2013 (17)) and in accordance with the WMO. Written informed consent will be obtained from all participants before study participation. Results of the study will be published in peer-reviewed scientific journals and will be presented at (inter)national conferences. If desired, participants will be informed about the outcomes of the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 years old
* ≥10 pack years of smoking
* primary diagnosis of COPD and post-bronchodilator ratio of forced expiratory volume in the first second (FEV1) to forced vital capacity (FVC) of less than 0.70.
* clinical indication for inpatient pulmonary rehabilitation in Ciro
* provided written informed consent

Exclusion Criteria:

* current, i.e. <12 months, (secondary) diagnosis of asthma according to the referring physician
* unstable concurrent cardiovascular, metabolic, renal, gastro-intestinal and musculoskeletal chronic diseases, as judged by the investigator
* chronic use of oral corticosteroids >10 mg prednisolone/day
* initiation of maintenance therapy with macrolides <6 weeks prior to study entry
* anemia, defined as hemoglobin level <8.1 mmol/L in men and <7.5 mmol/L in women
* participation in a study involving investigational or marketed products concomitantly or <8 weeks prior to study entry
* unable to read, speak or understand Dutch

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a primary diagnosis of COPD admitted for inpatient pulmonary rehabilitation at Ciro (Horn, The Netherlands).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory symptoms: EXACT | 8 weeks
  The EXAcerbations of Chronic pulmonary disease Tool (EXACT). The higher the score, the higher the disease burden. Scale: total score 0-100 points. Assessment: daily.
Respiratory symptoms: c-LRTI-VAS | 8 weeks
  The COPD- Lower Respiratory Tract Infection Visual Analogue Scales (c-LRTI-VAS). The higher the score, the higher the disease burden. Scale: 0-100 mm. Assessment: daily.
Vital signs: blood pressure | 8 weeks
  Systolic and diastolic blood pressure (mmHg). Assessment: daily.
Vital signs: heart rate | 8 weeks
  Heart rate (beats per minute). Assessment: daily.
Vital signs: oxygen saturation | 8 weeks
  Oxygen saturation (SpO2). Assessment: daily.
Vital signs: body temperature | 8 weeks
  Body temperature (degree Celsius). Assessment: daily.
Vital signs: breathing frequency | 8 weeks
  Breathing frequency (breaths per minute). Assessment: daily.
Pre-bronchodilator FEV1 | 8 weeks
  Absolute (L) and percentage of predicted (% pred) of the forced expiratory volume in 1 second (FEV1). Assessment: daily.
Pre-bronchodilator FVC | 8 weeks
  Absolute (L) and percentage of predicted (% pred) of the forced vital capacity (FVC). Assessment: daily.
Pre-bronchodilator PEF | 8 weeks
  Absolute (L/s) and percentage of predicted (% pred) of the peak expiratory flow (PEF). Assessment: daily.
Biomarkers: nasopharyngeal swabs | 8 weeks
  16S rRNA and ITS sequencing, and whole metatranscriptomic sequencing (WMTS). Assessment: enrollment, thrice-weekly (Monday-Wednesday-Friday) and exacerbation.
Biomarkers: venous blood | 8 weeks
  * SNP (associated with COPD, exacerbations and microbial infections) sequencing. Assessment: enrollment.
  * WMTS. Assessment: enrollment, exacerbation and outcome assessment.
  * ELISA-based multiplex cytokine analysis, anti-bacterial titer analysis, metabolomics, proteomics and WMTS. Assessment: enrollment, thrice-weekly (M-W-F), exacerbation and outcome assessment.
Biomarkers: spontaneous sputum | 8 weeks
  * 16S rRNA and ITS sequencing, WMTS, proteomics and metabolomics. Assessment: enrollment, thrice-weekly (M-W-F) and exacerbation.
  * Cell differentials and traditional bacterial culture at enrollment and exacerbation.
Biomarkers: stool | 8 weeks
  Whole metagenomic shotgun sequencing, and metabolomics. Assessment: enrollment, exacerbation, and outcome assessment.

SECONDARY OUTCOMES:
Basic characteristics | 8 weeks
  Age (years), sex (M/F), race (caucasian, negroid, asian), marital status (married/living together, divorced/separated, widow, single), smoking status (never smoked, ex-smoker, current smoker) and smoking history (pack years and type of tobacco), medical history and comorbidities (self- and physician reported), current medication use, chronic oxygen and non-invasive ventilation (L/min), as well as total number of moderate AECOPD and COPD-related hospitalizations in the previous 12 months, body length (m), body weight (kg), body mass index (BMI, kg/m2), fat free mass index (FFMI, kg/m2) and chest high-resolution computer tomography (HRCT) for post-hoc radiological quantification of pulmonary and extra-pulmonary features of COPD.
  These outcomes are aggregated to report the patient's overall basic characteristics.
  Assessment: enrollment.
Post-bronchodilator FEV1 | 8 weeks
  Absolute (L) and percentage of predicted (% pred) of the forced expiratory volume in 1 second (FEV1). Assessment: baseline and outcome assessment, as part of routine clinical care.
Post-bronchodilator FVC | 8 weeks
  Absolute (L) and percentage of predicted (% pred) of the forced vital capacity (FVC). Assessment: baseline and outcome assessment, as part of routine clinical care.
Post-bronchodilator PEF | 8 weeks
  Absolute (L/s) and percentage of predicted (% pred) of the peak expiratory flow (PEF). Assessment: baseline and outcome assessment, as part of routine clinical care.
Body plethysmography | 8 weeks
  Body plethysmography is performed to assess the absolute (L) and percentage of predicted (% pred) total lung capacity (TLC) and residual volume (RV), as well as the absolute (L/s) and percentage of predicted (% pred) intrathoracic gas volume (ITGV). Assessment: baseline assessment, as part of routine clinical care.
Diffusing capacity | 8 weeks
  The total (L) and % pred of the diffusing capacity (DLCO) and the DLCO per unit alveolar volume (KCO) are recorded. Additionally, DLCO and KCO will also be calculated corrected for hemoglobin. Assessment: baseline assessment, as part of routine clinical care.
Respiratory muscle strength | 8 weeks
  The absolute (cmH2O) and % pred maximal static inspiratory (MIP) and expiratory mouth pressures (MEP) are measured. Assessment: baseline assessment, as part of routine clinical care.
mMRC | 8 weeks
  The modified Medical Research Council (mMRC) is assessed to capture the severity of dyspnea. Scale: 0 to 4. Higher scores indicate a worse degree of dyspnea.
  Assessment: baseline and outcome assessment, as part of routine clinical care.
CAT | 8 weeks
  The COPD Assessment Test (CAT) is assessed to capture the health status. The total score ranges from 0 to 40 points, higher scores indicating a worse health status. Assessment: baseline and outcome assessment, as part of routine clinical care.
HADS | 8 weeks
  The Hospital Anxiety and Depression scale (HADS) questionnaire is assessed to indicate the level of anxiety and depression. Total scores for each subscale range from 0 (optimal) to 21 points (worst). A score of ≥10 points indicates the presence of symptoms of anxiety and depression. Assessment: baseline and outcome assessment, as part of routine clinical care.
Exercise capacity | 8 weeks
  The cardiopulmonary exercise test (CPET) is performed to capture the maximal exercise capacity (peak work rate [Wmax]). Assessment: baseline assessment.
  The constant work rate cycle test (CWRT) is performed to capture the submaximal work rate, 75% of the Wmax. Assessment: baseline and outcome assessment.
  The six-minute walk test (6MWT) is performed to capture the longest 6MWD for further analyses. Assessment: baseline and outcome assessment.
  These tests are performed as part of routine clinical care.
Muscle function | 8 weeks
  Muscle function will be determined through isometric and isokinetic quadriceps strength and endurance assessment. The highest peak torque will be determined (Nm) as well as the total amount of delivered work (J). Assessment: baseline and outcome assessment, as part of routine clinical care.
Hematology | 8 weeks
  Hemoglobin (mmol/L), hematocrit (L/L), thrombocytes (10E9/L), leukocytes (10E9/L), granulocytes (%), lymphocytes (10E9/L), lymphocytes (%), monocytes (%), eosinophilic granulocytes (10E9/L), eosinophilic granulocytes (%), basophilic granulocytes (%). Assessment: in venous blood at baseline and outcome assessment, as part of routine clinical care.
Chemistry | 8 weeks
  Glycated hemoglobin (HbA1c, mmol/mol and %), high density lipoprotein (HDL, mmol/L), low density lipoprotein (LDL, mmol/L), cholesterol (mmol/L), triglycerides (mmol/L), sodium (mmol/L), potassium (mmol/L), urea (mmol/L), creatinine (umol/L), aspartate aminotransferase (ASAT, U/L), alanine aminotransferase (ALAT, U/L), bilirubin (umol/L) and high sensitive C-reactive protein (hs-CRP, mg/L). Assessment: in venous blood at baseline and outcome assessment, as part of routine clinical care.
Arterial blood gas | 8 weeks
  An arterial blood sample is collected to determine the resting arterial partial pressure of oxygen (PaO2), carbon dioxide (PaCO2) and oxygen saturation (SpO2). Assessment: baseline assessment and at exacerbation, as part of routine clinical care.
Exacerbation markers | 8 weeks
  At exacerbation, as part of routine clinical care, venous blood is collected to determine the concentration of leukocytes (10E9/L), eosinophils (10E9/L), hs-CRP (mg/L), d-dimer (ug/L), NT-proBNP (pmol/L), troponin-T (ng/L).

CONTACTS AND LOCATIONS:
Overall Officials: Frits ME Franssen, Prof. Dr., Principal Investigator — Center of Expertise for Chronic Organ Failure
Locations (1):
- Ciro, Horn, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GOLD. Global strategy for the prevention, diagnosis and management of chronic obstructive pulmonary disease - 2022 report.
- [Background] Dransfield MT, Kunisaki KM, Strand MJ, Anzueto A, Bhatt SP, Bowler RP, Criner GJ, Curtis JL, Hanania NA, Nath H, Putcha N, Roark SE, Wan ES, Washko GR, Wells JM, Wendt CH, Make BJ; COPDGene Investigators. Acute Exacerbations and Lung Function Loss in Smokers with and without Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2017 Feb 1;195(3):324-330. doi: 10.1164/rccm.201605-1014OC. PMID 27556408
- [Background] Seemungal TA, Donaldson GC, Paul EA, Bestall JC, Jeffries DJ, Wedzicha JA. Effect of exacerbation on quality of life in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 May;157(5 Pt 1):1418-22. doi: 10.1164/ajrccm.157.5.9709032. PMID 9603117
- [Background] European Lung White Book: European Respiratory Society; 2003.
- [Background] CBS Doodsoorzakenstatistiek [Available from: www.cbs.nl.
- [Background] Wedzicha JA, Seemungal TA. COPD exacerbations: defining their cause and prevention. Lancet. 2007 Sep 1;370(9589):786-96. doi: 10.1016/S0140-6736(07)61382-8. PMID 17765528
- [Background] Vedel-Krogh S, Nielsen SF, Lange P, Vestbo J, Nordestgaard BG. Blood Eosinophils and Exacerbations in Chronic Obstructive Pulmonary Disease. The Copenhagen General Population Study. Am J Respir Crit Care Med. 2016 May 1;193(9):965-74. doi: 10.1164/rccm.201509-1869OC. PMID 26641631
- [Background] MacNee W, Donaldson K. Exacerbations of COPD: environmental mechanisms. Chest. 2000 May;117(5 Suppl 2):390S-7S. doi: 10.1378/chest.117.5_suppl_2.390s. PMID 10843983
- [Background] Viniol C, Vogelmeier CF. Exacerbations of COPD. Eur Respir Rev. 2018 Mar 14;27(147):170103. doi: 10.1183/16000617.0103-2017. Print 2018 Mar 31. PMID 29540496
- [Background] Hurst JR, Vestbo J, Anzueto A, Locantore N, Mullerova H, Tal-Singer R, Miller B, Lomas DA, Agusti A, Macnee W, Calverley P, Rennard S, Wouters EF, Wedzicha JA; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Susceptibility to exacerbation in chronic obstructive pulmonary disease. N Engl J Med. 2010 Sep 16;363(12):1128-38. doi: 10.1056/NEJMoa0909883. PMID 20843247
- [Background] Bafadhel M, McKenna S, Terry S, Mistry V, Reid C, Haldar P, McCormick M, Haldar K, Kebadze T, Duvoix A, Lindblad K, Patel H, Rugman P, Dodson P, Jenkins M, Saunders M, Newbold P, Green RH, Venge P, Lomas DA, Barer MR, Johnston SL, Pavord ID, Brightling CE. Acute exacerbations of chronic obstructive pulmonary disease: identification of biologic clusters and their biomarkers. Am J Respir Crit Care Med. 2011 Sep 15;184(6):662-71. doi: 10.1164/rccm.201104-0597OC. PMID 21680942
- [Background] Papi A, Bellettato CM, Braccioni F, Romagnoli M, Casolari P, Caramori G, Fabbri LM, Johnston SL. Infections and airway inflammation in chronic obstructive pulmonary disease severe exacerbations. Am J Respir Crit Care Med. 2006 May 15;173(10):1114-21. doi: 10.1164/rccm.200506-859OC. Epub 2006 Feb 16. PMID 16484677
- [Background] Wilkinson TMA, Aris E, Bourne S, Clarke SC, Peeters M, Pascal TG, Schoonbroodt S, Tuck AC, Kim V, Ostridge K, Staples KJ, Williams N, Williams A, Wootton S, Devaster JM; AERIS Study Group. A prospective, observational cohort study of the seasonal dynamics of airway pathogens in the aetiology of exacerbations in COPD. Thorax. 2017 Oct;72(10):919-927. doi: 10.1136/thoraxjnl-2016-209023. Epub 2017 Apr 21. PMID 28432209
- [Background] Dima E, Kyriakoudi A, Kaponi M, Vasileiadis I, Stamou P, Koutsoukou A, Koulouris NG, Rovina N. The lung microbiome dynamics between stability and exacerbation in chronic obstructive pulmonary disease (COPD): Current perspectives. Respir Med. 2019 Oct;157:1-6. doi: 10.1016/j.rmed.2019.08.012. Epub 2019 Aug 21. PMID 31450162
- [Background] Bouquet J, Tabor DE, Silver JS, Nair V, Tovchigrechko A, Griffin MP, Esser MT, Sellman BR, Jin H. Microbial burden and viral exacerbations in a longitudinal multicenter COPD cohort. Respir Res. 2020 Mar 30;21(1):77. doi: 10.1186/s12931-020-01340-0. PMID 32228581
- [Background] Braeken DCW, Spruit MA, Houben-Wilke S, Smid DE, Rohde GGU, Wouters EFM, Franssen FME. Impact of exacerbations on adherence and outcomes of pulmonary rehabilitation in patients with COPD. Respirology. 2017 Jul;22(5):942-949. doi: 10.1111/resp.12987. Epub 2017 Jan 31. PMID 28139873
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Derived] Waeijen-Smit K, DiGiandomenico A, Bonnell J, Ostridge K, Gehrmann U, Sellman BR, Kenny T, van Kuijk S, Peerlings D, Spruit MA, Simons SO, Houben-Wilke S, Franssen FME. Early diagnostic BioMARKers in exacerbations of chronic obstructive pulmonary disease: protocol of the exploratory, prospective, longitudinal, single-centre, observational MARKED study. BMJ Open. 2023 Mar 3;13(3):e068787. doi: 10.1136/bmjopen-2022-068787. PMID 36868599